CLINICAL TRIAL: NCT06142903
Title: THE COMPARATIVE EFFECTIVENESS OF 7 VERSUS 21 HOME-DELIVERED MEDICALLY TAILORED MEALS TO IMPROVE MALNUTRITION RISK IN MALNOURISHED PATIENTS WITH HEART FAILURE: A RANDOM ORDER CROSSOVER FEEDING TRIAL (MEDIMEALS)
Brief Title: Comparative Effectiveness of 7 Versus 21 Home-delivered Medically Tailored Meals to Improve Malnutrition Risk in Malnourished Patients With Heart Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 850914
Record Dates: First submitted 2023-11-15; First posted 2023-11-22 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Heart Failure; Malnutrition
Keywords: medically-tailored meals; diet quality; readmissions; emergency department visits
MeSH Terms: conditions — Heart Failure; Malnutrition

STUDY DESIGN:
Intervention Model Description: Consented patients will be randomized using a computer-generated scheme in REDcap to delivery of either 7 dinner meals or 21 meals (7 breakfast, 7 lunch, 7 dinner meals) each week for 4 weeks duration. At approximately day 0, 30 and 60 relative to discharge from the hospital, patients will be contacted by telephone to assess their malnutrition risk score, diet quality relative to AHA dietary goals, and obtain their self-measured weight and calf circumference.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 7 medically-tailored meals per week (Placebo Comparator): Patients will be randomized to medically tailored dinner meals delivered to their homes for four weeks.
  Interventions: Other: 7 versus 21 medically tailored meals per week
- 21 medically-tailored meals per week (Active Comparator): Patients will be randomized to three medically tailored dinner meals each day delivered to their homes for four weeks.
  Interventions: Other: 7 versus 21 medically tailored meals per week

INTERVENTIONS:
Other: 7 versus 21 medically tailored meals per week — Meals designed to support overall cardiovascular health will be provided to patients in their own home setting.

SUMMARY:
This protocol is designed to compare the effectiveness of two dietary intervention doses for patients with heart failure (HF) and malnutrition risk or malnutrition at hospital discharge. This random order crossover design will provide evidence as to whether the provision of dinner meals alone versus all 3 daily meals to patients' homes is more effective at improving malnutrition risk score, and secondarily unplanned emergency department visits and readmissions.

DETAILED DESCRIPTION:
1.1 Background and Relevant Literature Heart failure (HF) is a common clinical syndrome occurring in 6.2 million adults in the US with a cost of $30.7 million in 2012 due to health care services, medications, and missed days of work. The symptoms of HF result from the impaired ability of the heart to deliver blood and oxygen adequately to peripheral tissues.

Patients with HF at the Hospital of the University of Pennsylvania experience worse than expected clinical outcomes. Length of hospital stay in FY2021 (mean LOS 7.49 d, expected LOS 6.6 d) and FY22 (mean 7.21 d, expected 6.6 d), and 30-day readmissions were 17.1% in FY21 and 17.3% in FY22.

Malnutrition is a common comorbid condition with HF. In an observation of 4000 patients with HF, 57% had at least mild malnutrition, a condition that was associated with increased mortality. The malnutrition reported with HF comprises protein-energy malnutrition, muscle wasting, and cachexia, variables evaluated during malnutrition assessment.

Patients with malnutrition have worse clinical outcomes. Patients at our hospital who had moderate or severe disease-related malnutrition during the hospital stay had significantly more 30-day readmissions (40% versus 23%, OR 2.13, 1.82-2.48), greater mortality (OR 1.47, 1.0-1.99), and longer length of stay (15 vs 12 days, p= 0.0067) than patients who did not meet criteria for malnutrition4. In data from the 2012-2014 Nationwide Inpatient Sample, malnutrition was associated with mortality OR of 2.48, 2.3-2.66, almost double the admission cost, and longer length of stay of 8.7 days, 8.5-8.6 vs 5.3, 5.2-5.35.

The mainstay of HF disease management is patient self-management of medications, diet (restriction of Na with limited alcohol and fluid restriction to 1.5-2 L daily). Daily self-weighing is a strategy to detect fluid accumulation and permit adjustment of fluid intake or medical therapy. In addition to a Na restriction, the Diet Approach to Stop Hypertension or Mediterranean diet has been suggested. To optimize cardiovascular health and reduce cardiac deaths and strokes by 20%, the 2020 American Heart Association (AHA) guidelines included an evidence-based dietary approach targeting servings of six food groups (optimal intake of whole grains, fruits/vegetables, nuts/seeds/legumes, and fish; with limited intake of processed meats and sweet beverages)8 and with restriction of sodium intake to < 1500 mg and saturated fat to <7% of kcal. The DASH diet approach emphasizes intake of fruits, vegetables, whole grains, dairy, nuts/seeds/legumes, and limits intake of meat, sweets, and fats. A six-month nutrition intervention that included oral nutrition supplements in malnourished patients with HF significantly reduced mortality.

While readmissions in patients with HF are generally attributed to disease exacerbations, the disease exacerbations may be related to diet. Patients with HF should follow a strict Na-restricted heart healthy diet as a strategy to limit fluid accumulation that can exacerbate symptoms of edema, bloating and dyspnea. However, disease-related symptoms of fatigue or dyspnea may make preparing such a diet challenging because meals must be prepared without the use of processed or commercial frozen food items due to their high sodium and fat content.

Clinicians often treat patients with HF in the ED during emergency department visits (EDV) to avoid formal hospital admissions, though data on this outcome are not commonly reported. However, EDVs are disruptive to the quality of life of the patient and utilize hospital resources. We hypothesize that reducing malnutrition risk by providing medically-tailored meals may provide protection against 30-day unplanned readmissions and EDV.

Simple interventions such as provision of medically-tailored meals to the patient's home setting hold the potential to improve malnutrition and prevent both EDV and readmissions. One pilot trial compared 21 meals/week to standard care in patients with HF, with a trend towards fewer readmissions in the meals treatment arm. A small pilot in elderly patients, 38% of whom were diagnosed with HF, determined that it was feasible to provide 10 days of home-delivered meals, but lacked statistical power to determine the impact on readmissions by 45 days. However, there are no data to determine whether dinner meals alone will provide equivalent outcomes to 21 meals/week, or whether provision of medically tailored meals can improve malnutrition risk or reduce EDVs or readmissions.

2 Study Objectives The overall objective of the study is to determine whether the provision of 7 or 21 medically tailored meals per week to the patient in their home setting can improve malnutrition risk (MST score), and secondarily reduce 30-day unplanned EDV, readmissions, and improve diet quality by PDH score.

2.1 Primary Objective • To compare the effectiveness of home delivery of 7 versus 21 medically-tailored meals per week on improvement (reduction) in malnutrition risk (MST score).

2.2 Secondary Objectives

• To compare the effectiveness of home delivery of 7 versus 21 medically-tailored meals per week on unplanned 30-day EDV or readmissions and PHD score.

3 Investigational Plan Patients with HF who are identified with moderate or severe malnutrition during their HUP admission will be offered participation in the random order crossover design home-based feeding trial. Telephone visits with the patient at day 0±5, 30±5 and 60±5 will be used to gather MST, PHD, SARC-F, calf circumference, and weight data. The meals will be delivered weekly to the patient's home address by MANNA. The EDV and readmission outcomes will be adjudicated by the clinical dietitian in consultation with the cardiology medical team, as planned or unplanned events. Adverse events will be adjudicated for seriousness and relatedness to the diet intervention by Dr Bruce Kinosian, the study's safety officer.

3.1 General Design Consented patients will be randomized using a computer-generated scheme to delivery of either 7 dinner meals or 21 meals (7 breakfast, 7 lunch, 7 dinner meals) each week for 4 weeks duration. At approximately day 0, 30 and 60 relative to discharge from the hospital, patients will be contacted by telephone to assess their MST score, diet quality relative to AHA dietary goals, and obtain their self-measured weight and calf circumference.

3.2 Allocation to Interventional Group Subjects will be randomized in a one to one fashion to the order of 7 versus 21 meals/week intervention for one month followed immediately by the other treatment arm, using a computer-generated algorithm designed by the study statistician. MANNA contacts will be aware of the treatment arm assignment, but the study personnel will be blinded. Because the study meals are provided using the same foods, a washout period is not indicated.

3.3 Study Measures Each of the following tools will be collected by telephone contact with enrolled patients at approximately 0, 30 and 60 days relative to hospital discharge.

The Malnutrition Screening Tool (MST) score ranges from 0-5, with higher scores indicating greater risk of malnutrition.

The Penn Healthy Diet Survey (PHD) score ranges 0-64, with higher scores indicating a healthier diet.

Sarcopenia Screening Tool (SARC-F) score ranges 0-10 with higher results indicating greater debility.

Calf Circumference will be measured in cm by the patient or a caregiver at the maximum diameter of the calf using a paper measuring tape provided by the study prior to discharge.

Weight measured on the day of the telephone call will be recorded.

Adherence to medically-tailored meals will be determined by asking the patient how many of the meal entrees they were able to consume in the prior week.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* Diagnosis of Heart Failure (NYHA Class 1-3/ ACC/AHA Stage C) and moderate or severe malnutrition or malnutrition risk
* Residence within MANNA delivery area

Exclusion Criteria:

1. >90 years of age
2. Dementia/cognitive decline
3. Heart Failure stage 4 or D
4. Chronic kidney disease stage 5 or dialysis-dependent (GFR<30 mL/min/1.72 m2)
5. Unstable COPD as COPD flare within prior 3 months
6. Active cancer therapy
7. Pregnancy
8. Living in a residential facility such as prison, long-term care, rehabilitation, other
9. Allergy to foods on the menus
10. Persistent hyperkalemia (> 5 mEq/L) more than twice without excess potassium intake during hospital admission
11. Persistent hypotension (systolic BP<100 mm Hg) during the hospital admission
12. Systolic BP> 180 or diastolic BP >100 mmHg
13. Active substance or alcohol abuse

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
change in malnutrition risk | one month
  Malnutrition risk will be measured by the Malnutrition Risk Score survey

SECONDARY OUTCOMES:
Emergency Department Visits | one month
  ED visits will be evaluated relative to likelihood of dietary vs disease influence
Readmissions within 30 days | one month
  Readmissions during each 30-day window of diet treatment arm will be evaluated relative to the influence of diet versus disease

CONTACTS AND LOCATIONS:
Overall Officials: Charlene Compher, Principal Investigator — University of Pennsylvania
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
Data will not be shared.

REFERENCES:
- [Background] Compher CW, Quinn R, Haslam R, Bader E, Weaver J, Dudek S, Ritchie MD, Lewis JD, Wu GD. Penn Healthy Diet survey: pilot validation and scoring. Br J Nutr. 2024 Jan 14;131(1):156-162. doi: 10.1017/S0007114523001642. Epub 2023 Jul 31. PMID 37519237
- [Derived] Compher C, Henstenburg JA, Aloupis M, Sun A, Quinn R, Emery E, Thomas J, Crafford AG, Schwartz DR. The nutritional impact of 7 versus 21 home-delivered medically tailored meals in patients with heart failure and malnutrition risk: a random order crossover feeding trial (MEDIMEALS). BMC Nutr. 2025 Mar 18;11(1):56. doi: 10.1186/s40795-025-01036-y. PMID 40102963